CLINICAL TRIAL: NCT05938543
Title: Noninvasive Neuromodulation of a Novel Cerebellar Satiety Circuit in Prader-Willi Syndrome
Brief Title: Cerebellar TMS and Satiety in Prader-Willi Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Foundation for Prader-Willi Research (Other)
Responsible Party: Principal Investigator, Laura M Holsen, Associate Professor of Psychiatry, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2023P001354
Record Dates: First submitted 2023-06-13; First posted 2023-07-10 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Prader-Willi Syndrome
MeSH Terms: conditions — Prader-Willi Syndrome | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Active cerebellum rTMS (Experimental): Cerebellar targeted iTBS, once daily, one week
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — rTMS is a technique of TMS that allows for selective external manipulation of neural activity in a non-invasive manner. During rTMS a rapidly changing current is passed through an insulated coil placed against the scalp. This generates a temporary magnetic field, which in turn induces an electrical current in neurons and allows for modulation of neural circuitry.
  Other Name: iTBS

SUMMARY:
This study uses a noninvasive technique called transcranial magnetic stimulation (TMS) to study hyperphagia and satiety in Prader-Willi syndrome.

TMS is a noninvasive way of stimulating the brain, using a magnetic field to change activity in the brain. The magnetic field is produced by a coil that is held next to the scalp. In this study, the investigators will be stimulating the brain to learn more about how TMS might improve hyperphagia in Prader-Willi syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Prader-Willi syndrome

Exclusion Criteria:

* contraindications for TMS or MRI including :
* history of neurological disorder
* history of head trauma resulting in loss of consciousness
* history of seizures or diagnosis of epilepsy or first degree relative family history of epilepsy
* metal in brain or skull
* implanted devices such as a pacemaker, medication pump, nerve stimulator or ventriculoperitoneal shunt claustrophobic in MRI

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Retention of subjects in study assessments | 1-week post-TMS follow-up visit
  Retention of subjects for assessments at baseline and 1-week post-TMS follow-up visit, as measured by the percentage (%) of enrolled subjects who complete baseline assessments and then go on to complete the 1-week post-TMS follow-up visit.
Time required to enroll subjects into study | At study completion, up to 18 months
  Time required to enroll the target sample size (n=12) into the study
Change in BOLD response | baseline, 1-week post-TMS follow-up visit
  Change in functional activation of the cerebellum and ventral striatum will be assessed before (baseline) and after TMS stimulation (1-week post-TMS follow-up visit)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Holsen, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No